CLINICAL TRIAL: NCT02688751
Title: Contrast Enhanced Ultrasound Endoleak Detection Compared To Time-Resolved Computer Tomography Angiography in High Risk Endovascular Aneurysm Repair (EVAR) Surveillance Patients.
Brief Title: Contrast Enhanced Ultrasound, Endoleak Detection Following EVAR v1.3
Status: Completed | Type: Observational
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 5083; 15/NW/0908 (Other: NHS REC)
Record Dates: First submitted 2015-12-16; First posted 2016-02-23 (Estimated); Last update posted 2022-06-09 (Actual); Status verified 2016-09

CONDITIONS: Endoleak; Abdominal Aortic Aneurysm
MeSH Terms: conditions — Endoleak; Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: time-resolved CT Angiography — A multi-phase contrast CT
Procedure: Contrast Enhanced Ultrasound — A ultrasound scan with micro bubble contrast injection
  Other Names: CEUS

SUMMARY:
A single site cross-sectional comparison of paired diagnostic imaging modalities.

This study will show the sensitivity and specificity of CEUS in detecting the various types of endoleaks, in comparison to tCTA, following EVAR. It will collect data to allow comparison of diagnostic accuracy across modalities including CDU, CEUS and tCTA. It will collect time taken to perform the various types of scan, to allow healthcare costs to be calculated for each imaging modality.

DETAILED DESCRIPTION:
This study will show the sensitivity and specificity of CEUS in detecting the various types of endoleaks, in comparison to tCTA, following EVAR. It will collect data to allow comparison of diagnostic accuracy across modalities including CDU, CEUS and tCTA. It will collect time taken to perform the various types of scan, to allow healthcare costs to be calculated for each imaging modality.

Collected data will be analysed regarding two novel hypothesised methods of using CEUS information:

The first is recording temporal delay between contrast in graft and contrast in endoleak to define endoleak type. Potentially this could be used as a faster method of defining endoleak type in a surveillance programme.

The second is to identify/refute correlation between CEUS contrast to appear in endoleak vs tCTA contrast to appear in endoleak. If an association can be established, CEUS timings could potentially then be used to time 'standard' CTA phases to improve CTAs diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 or over
2. Able to give informed consent
3. Undergone an EVAR of infra-renal abdominal aortic aneurysm
4. Planned for CTA of EVAR

Exclusion Criteria:

1. Unable to receive CTA Contrast Allergy, Insufficient renal function for standard outpatient contrast study (eGFR <45) Overactive thyroid gland
2. Unable to receive CEUS contrast Previous reaction to Sonovue (Ultrasound Contrast) Allergy to sulphur hexafluoride (used in electrical industry in circuit breakers, switch gears & electrical equipment) Recent acute coronary syndrome or unstable angina, typical angina at rest or frequent or repeated angina/chest pain - all within previous 7 days Recent coronary intervention
3. Previous embolization of artery in region of EVAR (affects imaging quality)
4. BMI >30 (affects imaging quality)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients identified as being at increased risk of Type I/III endoleak following EVAR who require CTA & CEUS to confirm/refute this diagnosis.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2016-01-20 (Actual); Primary Completion 2018-03-20 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Ability to detect type I/III endoleak on CEUS as defined by presence/absence on tCTA | Immediate
  Will be presented as a Sensitivity & specificity

SECONDARY OUTCOMES:
Ability to detect type II endoleak on CEUS as defined by presence/absence on tCTA | Immediate
  Will be presented as a Sensitivity & specificity
Ability to predict secondary intervention on CEUS as defined by patients proceeding to secondary intervention | Immediate
  Will be presented as a Sensitivity & specificity
Confirm / refute association between temporal delay measured on CEUS and endoleak type as defined by tCTA, using the framework of general linear regression. | Immediate
  Temporal delay is the time difference between contrast arriving in the stent graft and contrast arriving in the endoleak on CEUS
Establish association between "CEUS contrast in endoleak" to "tCTA contrast in endoleak" by general linear regression analysis of timings recorded during CEUS & tCTA. | Immediate
Ability to predict secondary intervention of CDU, CEUS and tCTAas defined by patients proceeding to secondary intervention | 6 months
  Will be presented as a Sensitivity & specificity
Time taken for CDU, CEUS & tCTA scans to be performed as measured by observer. | Immediate
  Used to calculate total resource utilisation by individual scan types.

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasa R Vallabhaneni, MD, Study Chair — Liverpool University Hospitals NHS Foundation Trust
Locations (1):
- Royal Liverpool Hospital, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roy IN, Chan TY, Czanner G, Wallace S, Vallabhaneni SR. Prospective, single UK centre, comparative study of the predictive values of contrast-enhanced ultrasound compared to time-resolved CT angiography in the detection and characterisation of endoleaks in high-risk patients undergoing endovascular aneurysm repair surveillance: a protocol. BMJ Open. 2018 Apr 3;8(4):e020835. doi: 10.1136/bmjopen-2017-020835. PMID 29615450